CLINICAL TRIAL: NCT06295068
Title: Evaluation of the Aortic Regurgitation Index (ARi) Measured With the Opsens SavvyWire to Determine the Correlation Between Regurgitation Evaluation Using Echography and Aortography
Brief Title: Evaluation of ARi With OpSens SavvyWire
Acronym: ARi
Status: Terminated | Type: Observational
Why Stopped: Early termination.
Sponsor: Opsens, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PRT-1400-11
Record Dates: First submitted 2023-11-28; First posted 2024-03-06 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Aortic Valve Insufficiency
MeSH Terms: conditions — Aortic Valve Insufficiency | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Transcatheter Aortic Valve Replacement (TAVR) — Replacement of the aortic valve with use of the OpSens SavvyWire
Device: Balloon Aortic Valvuloplasty (BAV) — Dilation of the narrowed aortic valve by balloon inflation with use of the OpSens SavvyWire

SUMMARY:
The goal of this observational study is to establish the degree of agreement to Aortic Regurgitation (AR) severity during aortic valve intervention between the Aortic Regurgitation Index (ARi) measured by the Opsens SavvyWire, Echography and Aortography in subjects with severe aortic stenosis (AS) undergoing echo guided valve intervention. The main question it aims to answer is how the ARi measured with the Opsens SavvyWire compared with regurgitation evaluation derived by Echography and Aortography.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing TAVR suitable for intraoperative acquisition of TEE/TTE
* Age > 18 years
* Able and willing to give informed consent.

Exclusion Criteria:

* Hemodynamic instability making use of additional hemodynamic measurement inappropriate or 24-hour survival unlikely
* Subject is considered part of a vulnerable population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with severe aortic stenosis (AS) undergoing echo guided valve intervention
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Correlation of the Aortic Regurgitation Index (ARi) measured with the Opsens SavvyWire compared with regurgitation evaluation derived by Echography and Aortography | From the beginning of the procedure (first measurement is taken before the valve intervention) until to the end of the procedure (second measurement is taken after the valve Intervention), up to 2 hours

SECONDARY OUTCOMES:
Correlation of the Time Integration Aortic Regurgitation Index (TIARI) measured using the SavvyWire compare with regurgitation evaluation derived by Echography (TEE/TTE) and Aortography | From the beginning of the procedure (first measurement is taken before the valve intervention) until to the end of the procedure (second measurement is taken after the valve Intervention), up to 2 hours
Correlation of the Aortic Regurgitation Index Ratio measured using the Opsens SavvyWire compare with regurgitation evaluation derived by Echography and Aortography | From the beginning of the procedure (first measurement is taken before the valve intervention) until to the end of the procedure (second measurement is taken after the valve Intervention), up to 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Généreux, Dr, Principal Investigator — AHS Morristown Medical Center
Locations (1):
- AHS Morristown Medical Center, Morristown, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No